CLINICAL TRIAL: NCT06422507
Title: Multi-Center, Randomized, Double-Masked, Active-Controlled, Phase 3 Study of the Efficacy and Safety of 8 mg Aflibercept in Chinese Participants With Diabetic Macular Edema
Brief Title: A Study to Learn More About How Well 8 Milligram Aflibercept Works and How Safe it is in Chinese Participants With Diabetic Macular Edema
Acronym: PHOTONiC
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Bayer (Industry)
Collaborators: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 21583
Record Dates: First submitted 2024-05-15; First posted 2024-05-21 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: Diabetic Macular Edema
Keywords: DME
MeSH Terms: interventions — aflibercept; salicylhydroxamic acid

STUDY DESIGN:
Intervention Model Description: The study duration for a participant is approx 63 weeks. EOS is defined as the last visit of the last participant. HD aflibercept is the sponsor's study intervention under investigation. 322 participants will be randomized into 2 treatment groups in a ratio of 1:1 to receive either 2 mg aflibercept every 8 weeks following 5 initial monthly doses (2q8) or HD aflibercept (8mg) every 16 weeks following 3 initial monthly doses (HDq16). Randomization will be stratified according to baseline Central subfield thickness (CST <400µm, ≥400µm), baseline BCVA (<60 vs ≥60 ETDRS letters) and prior treatment for DME. Only 1 eye per participant is identified as the study eye. If a participant's fellow (non-study) eye has DME or Neovascular age-related macular degeneration (nAMD) that requires anti-Vascular endothelial growth factor (VEGF) treatment during the participant's involvement in the study, this eye should be treated with EYLEA (2mg aflibercept) and won't be considered an additional study eye.
Who Masked: Participant, Investigator
Masking Description: The study will be conducted in double-masked fashion. Study participants and masked study site personnel will remain masked to all randomization assignments throughout the study. The Sponsor personnel who are in regular contact with the study site will remain masked to all participant randomization assignments. The operational conduct of the study after the primary analysis at Week 48 will be maintained by a masked team. No decisions on data will be taken by any of the unmasked study personnel.
  To preserve masking, sham injections will be performed for all participants at treatment visits in which participants do not receive an active injection through Week 56.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- 2 mg aflibercept (Active Comparator): Participants that will be enrolled to this treatment arm will receive 2 mg aflibercept every 8 weeks following 5 initial monthly doses starting at Baseline (visit 2) (2q8) for the chosen "study eye". Randomization will be stratified according to baseline Central subfield thickness (CST) (<400 µm, ≥400 µm), baseline Best corrected visual acuity (BCVA) (<60 vs. ≥60 ETDRS letters) and prior treatment for DME.
  Interventions: Drug: 2 mg aflibercept (EYLEA, BAY 86-5321); Other: Sham
- 8 mg aflibercept (high dose) (Experimental): Participants that will be enrolled to this treatment arm will receive 8 mg (high dose - HD) aflibercept every 16 weeks following 3 initial monthly doses, starting at Baseline (Visit 2) (HDq16) for the chosen "study eye". Randomization will be stratified according to baseline Central subfield thickness (CST) (<400 µm, ≥400 µm), baseline Best corrected visual acuity (BCVA) (<60 vs. ≥60 ETDRS letters) and prior treatment for DME.
  Interventions: Drug: 8 mg aflibercept (BAY 86-5321) (High Dose); Other: Sham

INTERVENTIONS:
Drug: 8 mg aflibercept (BAY 86-5321) (High Dose) — High-dose (HD) aflibercept is the sponsor's study intervention under investigation. Dose formulation: solution in vial. Unit dose strength: 114.3 mg/mL, Dosage Level: 8 mg (70 µL), Route of Administration: Intravitreal (IVT) injection every 16 weeks following 3 initial monthly doses. Packaging/ Labeling: Study Intervention will be provided in sterile 3 mL glass vials. Each vial will be labeled as required per country requirement.
  Arms: 8 mg aflibercept (high dose)
Drug: 2 mg aflibercept (EYLEA, BAY 86-5321) — Aflibercept 2 mg is the sponsor's active comparator. Dose formulation: solution in vial. Unit dose strength: 40 mg/mL, Dosage Level: 2 mg (50 µL), Route of Administration: Intravitreal (IVT) injection every 8 weeks following 5 initial monthly doses. Packaging/ Labeling: Study Intervention will be provided in sterile 2 mL glass vials. Each vial will be labeled as required per country requirement. Aflibercept 2 mg for the non-study "fellow eye" treatment is considered an auxiliary medicinal product (AxMP) in this study. Fellow eye treatment will be allowed with 2 mg aflibercept, at the investigator's discretion for indications approved by governing authorities. The treated fellow eye will not be considered an additional study eye.
  Arms: 2 mg aflibercept
Other: Sham — To preserve masking, sham injections will be performed for all participants at treatment visits in which participants do not receive an active injection through Week 56. Sham kits will be assigned for visits requiring sham injections. The sham kits are empty but should be handled in the same way as the active study intervention kits.
  Sham injections will be given on visits when an active injection is not planned. During the study treatment period all participants will receive either an active injection (8 mg or 2 mg aflibercept) or a sham injection (for masking purposes) following their assigned treatment group and eligibility for Dose regimen modification (DRM).

SUMMARY:
Researchers are looking for a better way to treat people who have diabetic macular edema.

Diabetic macular edema (DME) is a diabetes-related eye disorder. In DME, the macula, which is the central part of the retina at the back of the eye, swells up resulting in vision problems. This happens due to leakage of fluid from damaged blood vessels.

The study treatment, 8 milligram (mg) aflibercept is injected into the eye. It works by blocking a protein called vascular endothelial growth factor (VEGF) which causes abnormal growth and leakage of blood vessels at the back of the eye.

A lower dose of aflibercept (2 mg) is already approved for the treatment of DME. Based on the findings of another study, the higher dose of aflibercept (8 mg) is expected to reduce the frequency of injections required for treating DME while being equally safe and working as well as the lower dose. The higher dose could make it easier to treat DME and improve quality of life for people with DME.

The main purpose of this study is to learn if high-dose (8 mg) aflibercept given every 16 weeks works as well as low-dose (2 mg) aflibercept given every 8 weeks in Chinese participants.

For this, the researchers will compare the change in participants' 'best corrected visual acuity' (BCVA) after 48 weeks of starting the treatment. BCVA is the clearest vision a participant can have with the help of corrective lenses, such as glasses. It will be measured by the number of letters the participant can read on an eye chart. This is known as their Early Treatment Diabetic Retinopathy Study (ETDRS) letter score.

Participants will be randomly (by chance) assigned to one of two treatment groups to receive study treatment as an injection into the eye up to Week 56:

* 2 mg aflibercept every 8 weeks after receiving 5 initial monthly doses
* 8 mg aflibercept every 16 weeks after receiving 3 initial monthly doses

Each participant will be in the study for around 63 weeks with up to 18 visits to the study site. This includes:

* one visit up to 21 days before the treatment starts during which the doctors will confirm that the participant can take part in the study
* 16 visits during which the treatment will be given. Most of these visits will have a gap of 4 weeks except for one visit that will happen a few days after the previous visit
* one visit 4 weeks after the treatment ends

During the study, the doctors and their study team will:

* check the participants' vision and their overall eye health using different eye tests
* check participants' health by performing tests such as blood and urine tests
* ask the participants questions about the disease and study treatment and how these impact their quality of life
* ask the participants what adverse events they are having An adverse event is any medical problem that a participant has during a study. Doctors keep track of all adverse events, irrespective of whether they think they are related to the study treatment.

Access to study treatment after the end of this study is not planned. Participants can switch to available approved treatments for DME.

DETAILED DESCRIPTION:
EYLEA (aflibercept 40 mg/mL solution for injection) at a dosage level of 2 mg administered intravitreally (IVT) is approved in over 100 countries for the treatment of DME. Despite the proven efficacy and safety of EYLEA in patients with DME, there remains an unmet need for alternative therapies that can decrease the burden of DME treatment via a reduction in the required frequency of IVT injections, while improving visual and anatomic outcomes. The overall one and two year results of PHOTON, a global phase 2/3 trial evaluating high dose (HD or 8 mg) aflibercept in participants with center-involved diabetic macular edema (DME), demonstrate the benefit of HD aflibercept for reducing the frequency of injections required for the treatment of DME while providing visual and anatomic outcomes non-inferior to and a safety profile indistinguishable from EYLEA, 2 mg aflibercept, the established standard of care for the treatment of DME. The observed reduction in the number of HD aflibercept injections required for the treatment of DME over 2 years in PHOTON is expected to translate into the benefit of reducing the burden of treatment and, thereby improving the quality of life for DME patients, their caregivers and health care providers. This study aims to investigate the efficacy and safety of HD aflibercept in Chinese participants with DME over 60 weeks with the primary objective of achieving non-inferior best corrected visual acuity (BCVA) with an extended dosing interval (every 16 weeks after 3 initial monthly injections) vs. 2 mg aflibercept (every 8 weeks after 5 initial monthly injections) similar to the results obtained in PHOTON. This study is designed to support the registration of HD aflibercept for the treatment of DME in China.

Primary Objective: The primary objective of the study is to determine if treatment with HD aflibercept at intervals of 16 weeks provides non-inferior best-corrected visual acuity (BCVA) compared to 2 mg aflibercept dosed every 8 weeks in Chinese participants

Secondary Objectives:

* To determine the effect of HD aflibercept vs. 2 mg aflibercept on anatomic and other visual measures of response;
* To evaluate the safety, immunogenicity and pharmacokinetics (PK) of HD aflibercept in Chinese participants.

Primary endpoint:

* Change from baseline in BCVA by ETDRS letter score at Week 48

Secondary endpoints:

* Change from baseline in BCVA by ETDRS letter score at Week 60
* Participants gaining ≥15 letters at Week 48 and Week 60
* Participants achieving an ETDRS letter score of at least 69 (approximate 20/40 Snellen equivalent) at Week 48
* Participants with no IRF and/or no SRF in the center subfield at Week 48
* Change from baseline in central subfield thickness (CST) at Week 48
* Change from baseline in leakage on fluorescein angiography (FA) at Week 48
* Change from baseline in National Eye Institute Visual Function Questionnaire (NEI-VFQ) total score at Week 48
* Occurrence of treatment-emergent adverse events (TEAEs) and serious adverse events (SAEs) through Weeks 48 and 60
* Participants developing a treatment-emergent ADA response or Nabs to aflibercept through EOS at Week 60
* Systemic exposure to aflibercept as assessed by plasma concentrations of free, adjusted bound, and total aflibercept from baseline through Week 48 This study is a phase 3, multi-center, randomized, double-masked, active-controlled study in Chinese participants with DME involving the center of the macula to investigate the efficacy and safety of HD aflibercept versus 2 mg aflibercept.

The primary objective of the study is to determine if treatment with HD aflibercept at 16 week intervals provides non-inferior BCVA compared to 2 mg aflibercept dosed every 8 weeks in Chinese participants.

322 eligible participants randomized in a 1:1 ratio to the following 2 treatment groups:

1. 2q8: 2 mg aflibercept every 8 weeks following 5 initial monthly doses (n=161) and
2. HDq16: HD aflibercept every 16 weeks following 3 initial monthly doses (n=161). The study consists of a screening period, a treatment period, and an end of study (EOS) visit at Week 60. The study duration for a participant is approximately 63 weeks. The EOS is defined as the last visit of the last participant. No study treatment will be administered at the EOS visit at Week 60.

HD aflibercept is the sponsor's study intervention under investigation. The following intervention groups are included in the study:

* 2 mg aflibercept every 8 weeks (2q8)
* 8 mg aflibercept every 16 weeks (HDq16)

ELIGIBILITY:
Key Inclusion Criteria:

* Men or women ≥18 years of age
* Chinese participants with type 1 or type 2 diabetes mellitus and diabetic macular edema (DME) with central involvement defined as CST ≥300 µm (or ≥320 µm on Heidelberg Spectralis) in the study eye as determined by the reading center at the screening visit and confirmed by the site at baseline visit
* BCVA early treatment diabetic retinopathy study (ETDRS) letter score of 78 to 24 (approximate Snellen equivalent of 20/32 to 20/320) in the study eye at the screening and baseline visits with decreased vision determined to be primarily the result of DME
* Women of childbearing potential (WOCBP) or men who are sexually active with partners of childbearing potential must agree to use highly effective contraception prior to the initial dose/start of the first treatment, during the study, and for at least 4 months after the last administration of study intervention.

Key Exclusion Criteria:

* Evidence of macular edema due to any cause other than diabetes mellitus in either eye
* Active proliferative diabetic retinopathy in the study eye
* Panretinal laser photocoagulation (PRP) or macular laser photocoagulation in the study eye within 12 weeks (84 days) of the screening visit
* IVT anti-VEGF treatment (aflibercept, ranibizumab, bevacizumab, conbercept, faricimab, brolucizumab, pegaptanib sodium) in the study eye within 12 weeks (84 days) of the screening visit
* Previous use of topical steroids within 4 weeks (28 days) of the screening visit or of intraocular or periocular corticosteroids in the study eye within 16 weeks (112 days) of the screening visit, or ILUVIEN or OZURDEX IVT implants at any time
* Prior ocular investigational agents (that have not been approved) in either eye (e.g., IVT, suprachoroidal injections, ocular implants, etc.) at any time.
* Previous treatment with an investigational or approved intraocular gene therapy or cell therapy in either eye at any time.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 333 (Actual)
Dates: Start 2024-05-29 (Actual); Primary Completion 2025-12-29 (Actual); Study Completion 2026-03-22 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in Best corrected visual acuity (BCVA) by Early Treatment Diabetic Retinopathy Study (ETDRS) letter score at Week 48 | Week 0 (Baseline) to Week 48
  The primary endpoint is the change from baseline in BCVA at Week 48. Efficacy analyses will be conducted using the Full analysis set (FAS).
  The primary efficacy analysis will be a comparison between 2 comparative arms: HDq16 vs. 2q8. The primary efficacy variable (Change from baseline in BCVA by ETDRS letter score at Week 48) will be analyzed using FAS with an Mixed Model for Repeated Measurements (MMRM) analysis model. The model includes baseline BCVA as a covariate, treatment group, baseline CST category, baseline BCVA category, prior DME treatment, and visit as fixed effects, and interaction terms for treatment by visit and baseline BCVA by visit. A Kenward-Roger approximation will be used for the denominator degrees of freedom.

SECONDARY OUTCOMES:
Change from baseline in BCVA by ETDRS letter score at Week 60 | Week 0 (Baseline) to Week 60
Participants gaining ≥15 letters at Week 48 and Week 60 | Week 48 and Week 60
Participants achieving an ETDRS letter score of at least 69 (approximate 20/40 Snellen equivalent) at Week 48 | Week 48
Participants with no Intraretinal fluid (IRF) and/or no Subretinal fluid (SRF) in the center subfield at Week 48 | Week 48
Change from baseline in central subfield thickness (CST) at Week 48 | Week 0 (Baseline) to Week 48
Change from baseline in leakage on fluorescein angiography (FA) at Week 48 | Week 0 (Baseline) to Week 48
Change from baseline in National Eye Institute Visual Function Questionnaire (NEI-VFQ) total score at Week 48 | Week 0 (Baseline) to Week 48
Occurrence of treatment-emergent adverse events (TEAEs) and serious adverse events (SAEs) through Weeks 48 and 60 | Week 48 to Week 60
Participants developing a treatment-emergent Anti-drug antibody (ADA) response or Nabs to aflibercept through EOS at Week 60 | Week 60
Systemic exposure to aflibercept as assessed by plasma concentrations of free, adjusted bound, and total aflibercept from baseline through Week 48 | Week 0 (Baseline) to Week 48

CONTACTS AND LOCATIONS:
Locations (52):
- China (50):
  - The Second Hospital of Anhui medical university, Hefei, Anhui
  - Beijing Hospital, Beijing, Beijing Municipality
  - Lanzhou University Second Hospital, Lanzhou, Gansu
  - Guangdong Provincial Hospital of TCM, Guangzhou, Guangdong
  - Guangzhou First People Hospital, Guangzhou, Guangdong
  - Zhujiang Hospital of Southern Medical University, Guangzhou, Guangdong
  - The People's Hospital of Guangxi Zhuang Autonomous Region, Nanning, Guangxi
  - The First Affiliated Hospital of Harbin Medical University, Harbin, Heilongjiang
  - Luoyang Third People's Hospital, Luoyang, Henan
  - Renmin Hosp., Wuhan Univ., Wuhan, Hubei
  - Nanjing First Hospital, Nanjing, Jiangsu
  - Affiliated hospital of Nantong university, Nantong, Jiangsu
  - The First Affiliated Hospital of NanChang University, Nanchang, Jiangxi
  - The Second Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - The Second Hospital of Jilin University, Changchun, Jilin
  - The First Hospital of Jilin University, Changchun, Jilin
  - Aier Eye Hospital (LIAONING), Shenyang, Liaoning
  - Shanxi Bethune Hospital, Taiyuan, Shanxi
  - Sichuan University West China Hospital, Chengdu, Sichuan
  - Taizhou Hospital of Zhejiang Province, Taizhou, Zhejiang
  - Zhengzhou Second People's Hospital, Erqi, Zhengzhou
  - Beijing Aier Intech Eye Hospital, Beijing
  - Beijing Friendship Hospital, Capital Medical University, Beijing
  - Capital Medical University (CMU) - Beijing Tongren Hospital, Beijing
  - Central South University - The Second Xiangya Hospital, Changsha
  - Chengdu Aier Ophthalmology Hospital, Chengdu
  - Chengdu University of Traditional Chinese Medicine - Teaching Hospital (Sichuan Province Traditional Chinese Medicine Hospital), Chengdu
  - The First Affiliated Hospital of Chongqing Medical Universit, Chongqing
  - Guangzhou Aier Ophthalmology Hospital, Guangzhou
  - Zhejiang University School of Medicine - The Second Affiliated Hospital, Hangzhou
  - Hebei eye hospital, Hebei
  - Henan Provincial Eye Hospital, Henan
  - Jinan Second People's Hospital, Jinan
  - Eye hospital of Shandong First Medical University, Jinan
  - People's Hospital of Ningxia Hui Autonomous Region - Opthalmology, Ningxia
  - Shandong University of Traditional Chinese Medicine Affiliated Ophthalmology Hospital, Shandong
  - Weifang Ophthalmology Hospital, Shandong
  - Shanghai eye disease prevention and control center, Shanghai
  - Shanghai General Hospital, Shanghai
  - Shanghai Jiao Tong University School of Medicine (SJTUSM) - XinHua Hospital, Shanghai
  - Eye & Ent Hospital of Fudan University, Shanghai
  - Joint Shantou International Eye Center (JSIEC)Shantou University & the Chinese University of Hong Kong, Shantou
  - Shanxi Eye Hospital, Shanxi
  - Shenyang He Eye Specialist Hospital, Shenyang
  - The Fourth People's Hospital of Shenyang, Shenyang
  - Shijiazhuang People's Hospital, Shijiazhuang
  - Tianjin Medical University Eye Hospital, Tianjin
  - Eye Hospital of Wenzhou Medical University, Wenzhou
  - Xi'an People's Hospital (Xi'an Fourth Hospital), Xi'an
  - Xianyang First People's Hospital, Xianyang
- Hong Kong (2):
  - Grantham Hospital, Hong Kong
  - Tseung Kwan O Hospital, Tseung Kwan O

IPD SHARING:
Plan to Share IPD: No
Availability of this study's data will later be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access. As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014.
  Interested researchers can use www.vivli.org to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the member section of the portal.

REFERENCES:
- See also: Click here to find further information and, after study completion, the study results according to Bayer's transparency standards. — https://clinicaltrials.bayer.com/study/21583